CLINICAL TRIAL: NCT04652999
Title: Relaxation Intervention in Patients With Diabetic Foot Ulcer: A Pilot Randomized Controlled Trial With a Nested Qualitative Study
Brief Title: Relaxation Intervention in Patients With Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Gabriela Ferreira, Master in Health Psychology, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEICVS015/2019
Record Dates: First submitted 2020-10-30; First posted 2020-12-04 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus; Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Relaxation; Ulcer Healing; Quality of Life; Pilot RCT
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Muscle Relaxation; Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: This is a Pilot Randomised Controlled Study of a Psychological Intervention (Eldridge et al., 2016; Grant et al., 2018). This study will use a mixed-methods approach nested in a pilot 3-arm randomized control design. Qualitative and quantitative data will be collected in order to provide better understanding about the feasibility and acceptability of the relaxation intervention in patients with DFU.
  Participants will be randomised at a ratio of 1:1 for the three conditions - EG, ACG and PCG; and will be evaluated on the day of the first chronic DFU appointment or nursing treatment (T0), two months later (at the end of the intervention in EG and ACG; T1), as well as six months later (T2) in a follow-up evaluation. Participants from all three groups will undergo standard treatment for the DFU, according to the guidelines of the Portuguese General Health Direction (DGS, 2010) and the International Working Group on the Diabetic Foot (IWGDF, 2015).
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible participants will be randomised into the three groups into blocks of variable size, multiples of three; and will be stratified according to: i) data collection site; ii) Chronic Renal Disease; and iii) Peripheral Arterial Disease; because they are factors of poor prognosis in the DFU healing (Ferreira et al., 2014). This procedure will be performed using an online random number generator, by a researcher external to the team involved in the implementation of this study, in order to ensure the concealment of the allocation of participants by the various groups (Pandis, 2012). After this procedure, it will not be possible to conceal the group to which the patient belongs from the researcher who will perform the psychological intervention. However, health professionals (doctors and nurses) will be blinded during the entire procedure, because they fill in the RESVECH 2.0, which assesses the DFU healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle Relaxation with Guided Imagery (Experimental): The participants in Experimental Group will receive four individual 45-minute sessions, every two weeks, of progressive muscle relaxation intervention with guided imagery focused on ulcer healing, carried out by the Psychologist responsible for implementing the project, on the day of the Diabetic Foot appointments.
  Interventions: Behavioral: Muscle Relaxation with Guided Imagery
- Active Control Group (Placebo Comparator): Participants in the Active Control Group will receive four individual 45-minute sessions of neutral guided imagery placebo, carried out by the Psychologist responsible for implementing the project, on the day of the Diabetic Foot appointments.
  Interventions: Behavioral: Neutral Guided Imagery
- Passive Control Group (No Intervention): The participants in the Passive Control Group will not receive any intervention nor placebo session.

INTERVENTIONS:
Behavioral: Muscle Relaxation with Guided Imagery — Relaxation intervention session begins with diaphragmatic breathing, followed by Jacobson's progressive muscle relaxation, which involves the contraction and subsequent relaxation of the 16 muscle groups of the body (forearm, arm, upper forehead, eye, mouth, jaw and throat, neck, shoulder, chest, stomach, thigh, leg and foot). The contraction is performed for 7 seconds while the relaxation lasts for about 40 to 50 seconds. The relaxation of the foot muscle group is only performed on the healthy foot, because dressing and bandages may bandage the foot with the DFU, which together with the typical joint stiffness of the diabetic foot, make it difficult to perform. After muscle relaxation, begins the guided imagery focused on DFU healing. The patient is instructed to think about his/her current state of health and to imagine the DFU as a dark area and the healing relaxation as a light associated to pleasant sensations, which will focus on the foot with DFU to heal it.
  Arms: Muscle Relaxation with Guided Imagery
Behavioral: Neutral Guided Imagery — This placebo consists on neutral guided imagery focused on themes of the patient's daily life before having DFU. Each session has a theme associated with the patient's life - family, work, friends and leisure. Initially, the patient is asked to think about an event related to the theme of the session of his/her choice, be it positive or negative, which occurred before patient has the current DFU. Then, questions are asked which allow a more detailed reconstruction of the event and the patient is asked to imagine according only to the instructions given. When the whole episode is remembered, the patient is asked to tell what he or she imagined/remembered in each of the questions given.
  Arms: Active Control Group

SUMMARY:
Diabetic foot ulcers (DFU) are one of the most serious complications of diabetes and can lead to amputations in 85% of cases, resulting in physical, psychological, family, social and economic consequences. Psychological interventions can contribute to the improvement of wound healing and, relaxation, in particular, seems to contribute to faster wound healing. More research is needed to assess the effectiveness of different types of intervention on different types of wounds, in particular on chronic wounds such as DFU.

This is a Pilot Randomised Controlled Study of a Psychological Intervention that aims to evaluate the feasibility and acceptability of a muscle relaxation intervention with guided imagery (experimental group - EG) compared to a neutral guided imagery placebo (active control group - ACG) and a group that does not receive any psychological intervention (passive control group - PCG), to inform a future definitive Randomised Controlled Study (RCT) that tests its effectiveness. This study will also examine, qualitatively, the perspectives of patients with DFU on the relaxation intervention, in order to check its acceptability and applicability; as well as the perspectives of health professionals on this adjuvant therapy, its applicability and integration into the care system of multidisciplinary diabetic foot consultations.

Participants have a diagnosis of Diabetes Mellitus and Diabetic Foot; one or two chronic ulcers active at the time of assessment; and clinical levels of stress or anxiety or depression. Participants will be randomized by the three conditions - EG, ACG and PCG - and assessed on the day of the first consultation or nursing treatment for chronic DFU (T0), two months later (T1), and six months later (T2; follow-up). Two weeks after T1, an interview will be conducted with patients with DFU that benefited from the relaxation sessions and to the health professionals who provided them the DFU care.

The results of the present study will contribute for a better understanding of DFU progression, healing, prevention of re-ulceration and future amputations and, consequently, for the improvement of patients' quality of life.

DETAILED DESCRIPTION:
General Aims:

This pilot RCT aims to assess the feasibility and acceptability of a muscle relaxation intervention with guided imagery (experimental group - GE) compared to a neutral guided imagery placebo (active control group - ACG) and a group that does not receive any psychological intervention (passive control group - PCG), prior to the implementation of a future definitive RCT that will assess its effectiveness.

This study will also examine, qualitatively, the perspectives of patients with DFU regarding the relaxation intervention, in order to check its acceptability and applicability; as well as the perspectives of health professionals on this adjuvant therapy, its applicability and integration into the multidisciplinary team of diabetic foot consultations.

Pilot RCT specific aims:

1. To evaluate the rates of eligibility, recruitment and adherence to the study protocol, participation in follow-up, and withdrawal. The degree of patient satisfaction with the relaxation intervention will also be assessed.
2. To verify the feasibility of the assessment protocol and to obtain preliminary estimates of the effects of the intervention on health outcome measures (degree of DFU healing, DFU-related quality of life, anxiety, depression and stress, DFU representations and physical and mental quality of life);
3. Synthesize the information to estimate the sample size required for a future definitive RCT.

   Qualitative study nested in Pilot RCT specific aims:
4. To understand the perspective of patients and health professionals about the relaxation sessions;
5. To explore the contribution of the relaxation sessions to the DFU healing and patients' quality of life;
6. To describe the changes perceived in the patient during the period of relaxation sessions;
7. To analyse the relevance of implementing relaxation sessions in the multidisciplinary team consultation of diabetic foot.

Data Analysis:

To assess the feasibility of this pilot study (aim 1), the rates of eligibility, recruitment and adherence to the study protocol, participation in the follow-up and withdrawal will be calculated and its results will be presented in percentage. The results of the degree of satisfaction with the intervention will be presented through mean and standard deviation. To obtain preliminary estimates of the intervention effects' on health outcome measures (aim 2), descriptive measures of the respective variables (means and standard deviations) will be calculated and Generalised Mixed Models will be used to check for statistically significant differences over time, in the different groups. Data will be analysed using IBM SPSS Statistics 26 for Mac. Finally, from the data obtained, the sample size for a future definitive RCT will be calculated (aim 3).

To answer the aims 4 to 7, a semi-structured interview guide consisting of open-ended questions will be administered to patients with DFU that benefited from the relaxation sessions and to the health professionals who provided them the DFU care. This script will remain unchanged throughout the interviews. The audio recording of the interviews will be done using a tablet, transcribed verbatim and anonymised in order to safeguard participants and data confidentiality. The transcripts of the interviews will be analysed in the same order as conducted, using the thematic content analysis technique (Bardin, 2016).

Sample size calculation:

The sample size calculation for a pilot RCT, considering the average effect size of 0.5, a statistical power of 80% and a significance level of 5%, revealed that 12 participants were needed in each of the groups (Cocks & Torgerson, 2013). This approach considers that a one-sided 80% confidence interval for the effect size will exclude the minimum clinically significant difference if the null hypothesis is true (Brown & Lilford, 2006).

Procedure:

The doctor or nurse, in the medical appointment, identifies patients that meet the medical inclusion criteria. Patients are invited to participate in the study by the Researcher at the end of the medical appointment and are informed about the aims of the study and the voluntary nature of participation through informed and informative consent. If patients agree to participate, they will sign the consent form. Nurses will then complete RESVECH 2.0 at the end of the appointment and doctors will complete the clinical questionnaire. Afterwards, the Researcher will accompany the patient to a room provided by the Hospital in order to administer the battery of questionnaires in the interview format.

After answering the questionnaires, the researcher will score the PSS and HADS instruments to identify the presence of significant clinical levels of stress, anxiety and depression, and if the patient is eligible, at the end of that week, the participant will be randomized into one of three possible groups.

In the next diabetic foot appointment, the respective participant will be informed about the group to which he or she has been allocated and whether will benefit, if appropriate, from four sessions of relaxation (EG) or neutral guided imagery (ACG), depending on the group. If the participant is available, the first session will take place on the same day. The following sessions will be scheduled according to the medical diabetic foot consultations. In each session, two assessments of blood pressure and heart rate will be performed, before starting the session and at the end of the session. At the end of the fourth session, the T1 assessment will be performed, with a new administration of the questionnaires. Six months after T0, the T2 (follow-up) evaluation will take place, with the last administration of the questionnaires.

The interviews with patients, who completed the four sessions of relaxation, and with health professionals, will be conducted two weeks after T1, by a different researcher than the one involved in the intervention, to reduce the bias of social desirability.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus diagnosis;
* Diagnosis of Diabetic Foot;
* Having one or two active chronic ulcers (> 6 weeks) at the time of the assessment;
* Being followed at the Multidisciplinary Consultation of the Diabetic Foot from the Centro Hospitalar Universitário do Porto (CHUP), at the Diabetic Foot Clinic from the Centro Hospitalar do Tâmega e Sousa (CHTS) and from the Hospital de Braga;
* Presenting clinical levels of stress (scores greater than 13 for males and greater than 17 for females on the Perceived Stress Scale) or anxiety or depression (scores greater than 11 on Hospital Anxiety and Depression Scale).

Exclusion Criteria:

* The active DFU at the time of the assessment being a relapse;
* Having more than two DFU currently active;
* Being on hemodialysis treatment;
* Presence of psychosis or dementia described in the patient's medical record;
* Having cancer disease;
* Having undergone a transplant;
* Receiving psychological counselling at the time of the assessment.

For the qualitative study nested in the Pilot RCT, participants must meet the same inclusion and exclusion criteria defined above, plus being allocated to the EG and have completed the four intervention sessions. From those participants, the following cases will be selected:

* Three typical cases of patients with neuropathic foot defined by the presence of neuropathic pain (e.g., heat, tingling, electrical shock), presence of distal pulses by palpation, and loss of protective sensitivity;
* Three typical cases of patients with neuroischemic foot defined by the presence of peripheral artery disease, intense-variable pain, absence of distal pulses by palpation, and variable protective sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of eligibility | Baseline (T0)
  This rate will result from the proportion between the number of eligible patients and the total number of observed patients, in percentage.
Rate of recruitment | Baseline (T0)
  This rate will result from the proportion between the number of patients who accepted to participate and the number of eligible patients, in percentage.
Rate of refusal | Baseline (T0)
  This rate will result from the proportion between the number of patients who rejected to participate in the study and the number of patients invited to participate, in percentage.
Rate of adherence to the study protocol | Through study completion, an average of 6 months
  This rate will result from the proportion between the number of patients who performed the assessments/intervention sessions and the number of patients who completed the baseline assessment (T0), in percentage.
Rate of participation in follow-up | Through study completion, an average of 6 months
  This rate will result from the proportion between the number of patients who participated in follow-up assessment and the number of patients who completed the baseline assessment (T0), presented in percentage.
Rate of dropout | Through study completion, an average of 6 months
  This rate will result from the proportion between the number of patients who dropout the study and the number of patients who completed the baseline assessment (T0), presented in percentage.
Patient satisfaction with the relaxation intervention | End of intervention/ 2 months later at post-test (T1)
  The degree of patients´ satisfaction with the relaxation intervention will be assessed through questions developed for this purpose, including the degree of general satisfaction with the sessions; the impact on stress, anxiety and depression, and wound healing after the four sessions; the degree of usefulness for patients with DFU; the desire to participate in future sessions; and the recommendation of the sessions to other patients with DFU. All the questions will be assessed on a Likert scale from 1 (very unsatisfied/ none/ totally disagree) to 5 (very satisfied/ extreme/ totally agree).

SECONDARY OUTCOMES:
Degree of DFU healing | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The degree of DFU healing will be assessed with the Portuguese version of "Resultados esperados de la valoración y evolución de la cicatrización de las heridas crónicas" Scale [Expected results of the evaluation and evolution of the healing of chronic wounds Scale - RESVECH 2.0] (Marques, 2015). The scores range from 0 to 35, where zero indicates complete healing.
Impact of DFU on patients' Quality of Life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The Diabetic Foot Ulcer Scale-Short Form (DFS-SF; Bann, Fehnel, & Gagnon, 2003; Research version by Pereira & Ferreira, 2018) will be used to assess patients´ DFU-related Quality of Life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better DFU-related quality of life.
Physical Quality of Life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The Short-Form Health Survey (SF-36; Ferreira, 1998; Ferreira, Ferreira, & Pereira, 2012) will be administered to assess patients' physical Health-related Quality of Life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better physical quality of life.
Mental Quality of Life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The Short-Form Health Survey (SF-36; Ferreira, 1998; Ferreira, Ferreira, & Pereira, 2012) will be administered to assess patients' mental Health-related Quality of Life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better mental quality of life.
Perceived Stress | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The overall stress perceived by the patient will be assessed through the Perceived Stress Scale (PSS; Trigo, Canudo, Branco, & Silva, 2010).
  Scores range between 0 and 40, with higher results indicating higher levels of perceived stress.
Emotional Distress | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The emotional distress will be assessed through the total score of the Hospital Anxiety and Depression Scale, comprising both anxiety and depression scales (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 42, with higher results indicating higher levels of distress.
Anxiety symptoms | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The anxious symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of anxiety symptoms.
Depression symptoms | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The depressive symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of depression symptoms.
Adherence to DFU Care | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  Patient adherence to DFU care will be assessed through the DFU Care Adherence Questionnaire (Research Version by Pereira, Dantas, Brandão, Santos, Carvalho, & Ferreira, 2018), which was developed for this study, according to the guidelines of the Portuguese General Direction of Health (DGS, 2010) and the International Working Group on the Diabetic Foot (IWGDF, 2015). Higher scores indicate better adherence to DFU care.
Representations regarding the DFU | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  Patient representations regarding the DFU will be evaluated through the Illness Perception Questionnaire - Brief (IPQ-B; Figueiras et al., 2010). The response scale ranges from 0 to 10. Higher scores indicate more threatening representations regarding DFU.
Systolic Pressure | Before and after each intervention (EG) or placebo (ACG) at 2 weeks (1st Session), 4 weeks (2nd Session), 6 weeks (3rd Session) and 8 weeks (4th Session), after the baseline (T0)
  Systolic pressure in millimeters of mercury (mmHg) will be assessed through a validated and certified blood pressure measuring device.
Diastolic Pressure | Before and after each intervention (EG) or placebo (ACG) at 2 weeks (1st Session), 4 weeks (2nd Session), 6 weeks (3rd Session) and 8 weeks (4th Session), after the baseline (T0)
  Diastolic pressure in millimeters of mercury (mmHg) will be assessed through a validated and certified blood pressure measuring device.
Heart rate | Before and after each intervention (EG) or placebo (ACG) at 2 weeks (1st Session), 4 weeks (2nd Session), 6 weeks (3rd Session) and 8 weeks (4th Session), after the baseline (T0)
  Heart rate in beats per minute (bpm) will be assessed through a validated and certified blood pressure measuring device.

OTHER OUTCOMES:
Sociodemographic Data | Baseline (T0)
  The following socio-demographic data will be collected: gender; age; living environment; marital status; professional status; monthly income; if there is an informal caregiver, what is the degree of kinship with the caregiver and the quality of the patient's relationship with the caregiver; as well as some questions regarding access to health care.
Health Literacy | Baseline (T0)
  The level of health literacy will be assessed through the Medical Term Recognition Test (METER; Paiva et al., 2014).
Clinical Data | Baseline (T0), end of intervention/ 2 months later at post-test (T1), and after a six month follow-up (T2)
  The clinical data collected through a clinical questionnaire developed for this study will be: alcohol and tobacco consumption, presence and intensity of ulcer-related pain, and other symptomatic foot complaints; the type and duration of diabetes, HbA1c levels, duration of diabetic foot ulcer, type of foot and type of ulcer (PEDIS classification), location of the ulcer, recognised complications and comorbidities, type of treatment provided at the consultation, number of medical and nursing visits, date of DFU healing, and appearance of new ulcers. Psychophysiological parameters such as transcutaneous O2 pressure (TCPO2) where appropriate; blood pressure and heart rate; will also be assessed, the latter two being evaluated by an automatic blood pressure measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Ferreira, Master, Principal Investigator — School of Psychology, University of Minho; M.Graça Pereira, PhD, Study Director — School of Psychology, University of Minho
Locations (2):
- Portugal (2):
  - Clínica do Pé Diabético, Centro Hospitalar do Tâmega e Sousa, Penafiel
  - Centro Hospitalar Universitário do Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bann CM, Fehnel SE, Gagnon DD. Development and validation of the Diabetic Foot Ulcer Scale-short form (DFS-SF). Pharmacoeconomics. 2003;21(17):1277-90. doi: 10.2165/00019053-200321170-00004. PMID 14986739
- [Background] Bardin L. Análise de Conteúdo [Content Analysis]. 2016; São Paulo, Brasil: Almedina. Brasil.
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Direção-Geral de Saúde, DGS [General Health Direction, Portugal] Circular Normativa Nº:05/PNPCD: Pé Diabético, Programa Nacional de Prevenção e Controlo da Diabetes (PNPCD) [Normative Circular Nº: 05 / PNPCD: Diabetic Foot, National Diabetes Prevention and Control Program]; 2010. Retrieved from http://www.dgs.pt/?cr=15718
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Ferreira P. A medição do estado de saúde: Criação da versão portuguesa do MOS SF-36 [Measuring health status: Creation of the Portuguese version of MOS SF-36]. Coimbra: Centro de Estudos e Investigação em Saúde, Faculdade de Economia, Universidade de Coimbra; 1998.
- [Background] Ferreira PL, Ferreira LN, Pereira LN. Medidas sumário física e mental de estado de saúde para a população portuguesa [Physical and mental summary measures of health state for the Portuguese population]. Revista Portuguesa de Saúde Pública. 2012;30(2):163-171. doi:10.1016/j.rpsp.2012.12.007.
- [Background] Ferreira V, Martins J, Loureiro L, Loureiro T, Borges L, Silveira D, … Almeida R. Consulta multidisciplinar do pé diabético: Avaliação dos fatores de mau prognóstico [Multidisciplinary consultation of diabetic foot - factors related with bad prognosis]. Angiologia e Cirurgia Vascular. 2014;10:146-150. doi:10.1016/j.ancv.2014.08.005
- [Background] Figueiras M, Marcelino DS, Claudino A, Cortes MA, Maroco J, Weinman J. Patients' illness schemata of hypertension: the role of beliefs for the choice of treatment. Psychol Health. 2010 Apr;25(4):507-17. doi: 10.1080/08870440802578961. PMID 20204931
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] International Working Group on the Diabetic Foot [IWGDF] International Consensus on the Diabetic Foot. International Diabetes Foundation; 2015. Retrieved from http://www.iwgdf.org/files/2015/website_prevention.pdf
- [Background] Marques JM. Adaptação cultural e validação para a população portuguesa de um instrumento de monitorização de feridas crónicas - escala RESVECH 2.0 [Cultural adaptation and validation for the Portuguese population of a chronic wound monitoring instrument - RESVECH 2.0 scale] (Master's Thesis). Instituto de Ciências da Saúde da Universidade Católica, Porto; 2015.
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Paiva D, Silva S, Severo M, Ferreira P, Santos O, Lunet N, Azevedo A. Cross-cultural adaptation and validation of the health literacy assessment tool METER in the Portuguese adult population. Patient Educ Couns. 2014 Nov;97(2):269-75. doi: 10.1016/j.pec.2014.07.024. Epub 2014 Jul 22. PMID 25107513
- [Background] Pandis N. Randomization. Part 3: allocation concealment and randomization implementation. Am J Orthod Dentofacial Orthop. 2012 Jan;141(1):126-8. doi: 10.1016/j.ajodo.2011.09.003. No abstract available. PMID 22196195
- [Background] Trigo M, Canudo N, Branco F, Silva D. Estudo das propriedades psicométricas da Perceived Stress Scale (PSS) na população Portuguesa [Psychometric proprieties of the Perceived Stress Scale (PSS) in Portuguese population]. Psychologica. 2010;53:353-378. doi:10.14195/1647-8606_53_17
- [Derived] Ferreira G, Bernardo AC, Carvalho A, Pereira MG. Relax to Heal? Perspectives of Patients with Diabetic Foot Ulcers and Health Professionals on Relaxation Sessions for Wound Healing. Adv Skin Wound Care. 2023 Jun 1;36(6):1-10. doi: 10.1097/01.ASW.0000922832.62539.a3. Epub 2023 Apr 4. PMID 37017401